CLINICAL TRIAL: NCT01193725
Title: Comparing Virtual Reality Exposure Therapy to Prolonged Exposure in the Treatment of Soldiers With PTSD
Brief Title: Exposure Therapy for Active Duty Soldiers With Post Traumatic Stress Disorder
Acronym: VRPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Telehealth and Technology (U.S. Federal Agency)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDO-09-8014; W81XWH-08-2-0015 (Other Grant/Funding Number: UA Army MRMC)
Record Dates: First submitted 2010-08-30; First posted 2010-09-02 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Stress Disorders, Post Traumatic
Keywords: Combat Disorders; Exposure Therapy; Army Personnel
MeSH Terms: conditions — Combat Disorders | interventions — Virtual Reality Exposure Therapy; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prolonged Exposure Therapy (PE) (Active Comparator): The PE protocol is based on manualized procedures, which are derived from the theory that effective treatment for PTSD requires that the underlying pathological fear structure be activated and paired with new information that is incompatible with the fear structure. PE involves imaginal exposure and in vivo exposure as the two primary strategies to elicit repeated confrontation of feared but objectively safe thoughts, feelings, situations and events.
  Interventions: Behavioral: Prolonged Exposure Therapy (PE)
- Virtual Reality Exposure Therapy (VRET) (Experimental): The VRET protocol follows the same procedures as the PE protocol with the primary exception being that all instances of imaginal exposure will be augmented by immersion into Virtual Iraq environments, thus creating a situation known as immersive exposure.
  Interventions: Behavioral: Virtual Reality Exposure Therapy (VRET)
- Waitlist (Placebo Comparator): The waitlist (WL) participants will be asked to refrain from psychotherapy during the 5 weeks of study participation.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy (PE) — Prolonged exposure therapy will consist of 10 treatment sessions lasting 90 - 120 minutes each, with additional between-session homework assignments.
  Other Names: PE
  Arms: Prolonged Exposure Therapy (PE)
Behavioral: Virtual Reality Exposure Therapy (VRET) — Virtual Reality Exposure Therapy will consist of 10 treatment sessions lasting 90 -120 minutes with additional between-session homework assignments.
  Other Names: VRE; VRET
  Arms: Virtual Reality Exposure Therapy (VRET)
Behavioral: Waitlist — This group will refrain from psychotherapy until after the completion of the 5 weeks of study participation
  Other Names: WL; Waitlist Control Group
  Arms: Waitlist

SUMMARY:
This study is evaluating the efficacy of virtual realty exposure therapy (VRET)by comparing it to prolonged exposure therapy (PE) and a waitlist (WL) group for the treatment of post traumatic stress disorder (PTSD) in active duty (AD) Soldiers with combat-related trauma. The investigators will test the general hypotheses that 10 sessions of VRET or PE will successfully treat PTSD, therapeutically affect levels of physiological arousal, and significantly reduce perceptions of stigma toward seeking behavioral health services.

DETAILED DESCRIPTION:
The rationale for this study is based on growing evidence demonstrating that VRET is an efficacious treatment for PTSD and holds the potential to improve access to care for Soldiers who would otherwise avoid treatment. Although PE is considered one of the most effective cognitive-behavioral therapies (CBT) for treatments for PTSD, there are reasons why it may not be the most viable option for many Soldiers. First, Prolonged exposure requires a level of emotional engagement during exposure to the trauma that many patients are unable to obtain. Second, stigma and concerns about how Soldiers will be perceived by peers and leadership has a dramatic impact on whether a Soldier will seek care. VRET may address these concerns and may also improve treatment outcomes and access to care by augmenting the patient's re-living of the trauma with a sensory-rich environment and moderating stigma perceptions by offering non-traditional treatment that is a preferable option for many Soldiers who are reluctant to seek out traditional talk therapies. Despite its promise as a viable treatment option, few studies have examined VRET for combat-related PTSD and there are no published studies that have compared VRET to PE in the treatment of combat-related PTSD. Positive results may provide new treatment options for all Soldiers, but should prove to be an especially attractive option for Soldiers who either do not respond to, or are reluctant to engage in other established therapies such as PE.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis as assessed by CAPS
* history of deployment in support of OIF/OEF
* non sexually based deployment related trauma
* three or more months since index trauma
* stable on psychotropic medications for 30 days

Exclusion Criteria:

* index trauma in the last three months
* history of schizophrenia, other psychotic or bipolar disorder
* history of organic brain disorder
* suicidal risk or intent or self-mutilating behavior requiring hospitalization in the last 6 months
* ongoing threatening situation
* current drug or alcohol dependence
* history of seizures
* prior history of PE for PTSD
* other current psychotherapy
* physical condition that interferes with proper use of Virtual Reality head mounted display
* history of loss of consciousness since entering active duty service greater than 15 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-03; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS) | Screening Visit ( Day 1)
  The CAPS is a structured interview that assesses all DSM-IV PTSD criteria in terms of frequency and intensity. Scores are computed for Intrusion, Avoidance and Hyperarousal symptom clusters, as well as a Total score.
Clinician-Administered PTSD Scale (CAPS) | 2.5 weeks (or after treatment session 5)
  The CAPS is a structured interview that assesses all DSM-IV PTSD criteria in terms of frequency and intensity. Scores are computed for Intrusion, Avoidance and Hyperarousal symptom clusters, as well as a Total score.
Clinician-Administered PTSD Scale (CAPS) | 5 weeks (or after treatment session 10)
  The CAPS is a structured interview that assesses all DSM-IV PTSD criteria in terms of frequency and intensity. Scores are computed for Intrusion, Avoidance and Hyperarousal symptom clusters, as well as a Total score.
Clinician-Administered PTSD Scale (CAPS) | 12 Week follow-up
  The CAPS is a structured interview that assesses all DSM-IV PTSD criteria in terms of frequency and intensity. Scores are computed for Intrusion, Avoidance and Hyperarousal symptom clusters, as well as a Total score.
Clinician-Administered PTSD Scale (CAPS) | 26 Week follow-up
  The CAPS is a structured interview that assesses all DSM-IV PTSD criteria in terms of frequency and intensity. Scores are computed for Intrusion, Avoidance and Hyperarousal symptom clusters, as well as a Total score.

SECONDARY OUTCOMES:
PTSD Checklist (PCL-C) | Screening Visit (Day 1)
  The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
Primary Care PTSD Screen (PC-PTSD) | Screening Visit(Day 1)
  The PC-PTSD is a four-item measure designed to screen for PTSD.
Beck Depression Inventory-II (BDI-II) | Screening Visit(Day 1)
  This self report measure of depression contains 21 items that are rated on a 4 point scale.
Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS) | Screening Visit(Day 1)
  The IASMHS is a 24 item assessment of help-seeking attitudes. It includes the following three factors based on components of Ajzen's Theory of Planned Behavior: Psychological Openness, Help-seeking Propensity and Indifference to Stigma.
Perceived Stigma Measure (PSS) | Screening Visit(Day 1)
  Stigma will be measured using a 5 question assessment scale.
Suicide Risk Assessment | Screening Visit(Day 1)
  Due to the nature of the questions, this is deemed to be of safety nature.
Beck Anxiety Inventory (BAI) | Screening Visit(Day 1)
  The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
BASIS-24 | Screening Visit(Day 1)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
Subjective Units of Distress (SUDs) | Treatment session 1 (week 1)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Side Effects Questionnaire | Treatment session 1(week 1)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
PTSD Checklist (PCL-C) | 2.5 weeks (or after treatment session 5)
  The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
PTSD Checklist (PCL-C) | 5 weeks (or after treatment session 10)
  The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
PTSD Checklist (PCL-C) | 12 Week Follow-up
  The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
PTSD Checklist (PCL-C) | 26 Week Follow-up
  The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
Primary Care PTSD Screen (PC-PTSD) | 2.5 weeks (or after treatment session 5)
  The PC-PTSD is a four-item measure designed to screen for PTSD.
Primary Care PTSD Screen (PC-PTSD) | 5 weeks (or after treatment session 10)
  The PC-PTSD is a four-item measure designed to screen for PTSD.
Primary Care PTSD Screen (PC-PTSD) | 12 Week Follow-up
  The PC-PTSD is a four-item measure designed to screen for PTSD.
Primary Care PTSD Screen (PC-PTSD) | 26 Week Follow-up
  The PC-PTSD is a four-item measure designed to screen for PTSD.
Beck Depression Inventory-II (BDI-II) | 2.5 weeks (or after treatment session 5)
  This self report measure of depression contains 21 items that are rated on a 4 point scale.
Beck Depression Inventory-II (BDI-II) | 5 weeks (or after treatment session 10)
  This self report measure of depression contains 21 items that are rated on a 4 point scale.
Beck Depression Inventory-II (BDI-II) | 12 Week Follow-up
  This self report measure of depression contains 21 items that are rated on a 4 point scale.
Beck Depression Inventory-II (BDI-II) | 26 Week Follow-up
  This self report measure of depression contains 21 items that are rated on a 4 point scale.
Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS) | 2.5 weeks (or after treatment session 5)
  The IASMHS is a 24 item assessment of help-seeking attitudes. It includes the following three factors based on components of Ajzen's Theory of Planned Behavior: Psychological Openness, Help-seeking Propensity and Indifference to Stigma.
Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS) | 5 weeks (or after treatment session 10)
  The IASMHS is a 24 item assessment of help-seeking attitudes. It includes the following three factors based on components of Ajzen's Theory of Planned Behavior: Psychological Openness, Help-seeking Propensity and Indifference to Stigma.
Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS) | 12 Week Follow-up
  The IASMHS is a 24 item assessment of help-seeking attitudes. It includes the following three factors based on components of Ajzen's Theory of Planned Behavior: Psychological Openness, Help-seeking Propensity and Indifference to Stigma.
Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS) | 26 Week Follow-up
  The IASMHS is a 24 item assessment of help-seeking attitudes. It includes the following three factors based on components of Ajzen's Theory of Planned Behavior: Psychological Openness, Help-seeking Propensity and Indifference to Stigma.
Perceived Stigma Measure (PSS) | 2.5 weeks (or after treatment session 5)
  Stigma will be measured using a 5 question assessment scale.
Perceived Stigma Measure (PSS) | 5 weeks (or after treatment session 10)
  Stigma will be measured using a 5 question assessment scale.
Perceived Stigma Measure (PSS) | 12 Week Follow-up
  Stigma will be measured using a 5 question assessment scale.
Perceived Stigma Measure (PSS) | 26 Week Follow-up
  Stigma will be measured using a 5 question assessment scale.
Suicide Risk Assessment | 2.5 weeks (or after treatment session 5)
  Due to the nature of the questions, this is deemed to be of safety nature.
Suicide Risk Assessment | 5 weeks (or after treatment session 10)
  Due to the nature of the questions, this is deemed to be of safety nature.
Suicide Risk Assessment | 12 Week Follow-up
  Due to the nature of the questions, this is deemed to be of safety nature.
Suicide Risk Assessment | 26 Week Follow-up
  Due to the nature of the questions, this is deemed to be of safety nature.
Beck Anxiety Inventory (BAI) | 2.5 weeks (or after treatment session 5)
  The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
Beck Anxiety Inventory (BAI) | 5 weeks (or after treatment session 10)
  The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
Beck Anxiety Inventory (BAI) | 12 Week Follow-up
  The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
Beck Anxiety Inventory (BAI) | 26 Week Follow-up
  The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
BASIS-24 | Treatment session 1(week 1)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | Treatment session 2(week 1)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | Treatment session 3 (Week 2)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | Treatment session 4(Week 2)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | Treatment session 5 (Week 2.5)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | Treatment session 6 (Week 3)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | Treatment session 7 (Week 4)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | Treatment session 8 (Week 4)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | Treatment session 9 (Week 5)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | Treatment session 10 (Week 5)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | 2.5 weeks (or after treatment session 5)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | 5 weeks (or after treatment session 10)
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | 12 Week Follow-up
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
BASIS-24 | 26 Week Follow-up
  To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
Subjective Units of Distress (SUDs) | Treatment session 2(week 1)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Subjective Units of Distress (SUDs) | Treatment session 3(Week 2)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Subjective Units of Distress (SUDs) | Treatment session 4(Week 2)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Subjective Units of Distress (SUDs) | Treatment session 5 (Week 2.5)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Subjective Units of Distress (SUDs) | Treatment session 6 (Week 3)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Subjective Units of Distress (SUDs) | Treatment session 7 (Week 4)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Subjective Units of Distress (SUDs) | Treatment session 8 (Week 4)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Subjective Units of Distress (SUDs) | Treatment session 9 (Week 5)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Subjective Units of Distress (SUDs) | Treatment session 10 (Week 5)
  Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Side Effects Questionnaire | Treatment session 2(week 1)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
Side Effects Questionnaire | Treatment session 3(Week 2)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
Side Effects Questionnaire | Treatment session 4(Week 2)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
Side Effects Questionnaire | Treatment session 5(Week 2.5)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
Side Effects Questionnaire | Treatment session 6 (Week 3)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
Side Effects Questionnaire | Treatment session 7 (Week 4)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
Side Effects Questionnaire | Treatment session 8 (Week 4)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
Side Effects Questionnaire | Treatment session 9 (Week 5)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
Side Effects Questionnaire | Treatment session 10 (Week 5)
  The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Gahm, PhD, Principal Investigator — DCoE - National Center for Telehealth and Technology; Greg Reger, PhD, Principal Investigator — DCoE - National Center for Telehealth and Technology
Locations (1):
- National Center for Telehealth and Technology, Tacoma, Washington, United States

REFERENCES:
- [Background] Rothbaum BO, Hodges LF. The use of virtual reality exposure in the treatment of anxiety disorders. Behav Modif. 1999 Oct;23(4):507-25. doi: 10.1177/0145445599234001. PMID 10533438
- [Background] Pole N. The psychophysiology of posttraumatic stress disorder: a meta-analysis. Psychol Bull. 2007 Sep;133(5):725-46. doi: 10.1037/0033-2909.133.5.725. PMID 17723027
- [Background] Jaycox LH, Foa EB, Morral AR. Influence of emotional engagement and habituation on exposure therapy for PTSD. J Consult Clin Psychol. 1998 Feb;66(1):185-92. doi: 10.1037//0022-006x.66.1.185. PMID 9489273
- [Background] Difede J, Cukor J, Patt I, Giosan C, Hoffman H. The application of virtual reality to the treatment of PTSD following the WTC attack. Ann N Y Acad Sci. 2006 Jul;1071:500-1. doi: 10.1196/annals.1364.052. PMID 16891607
- [Background] Rothbaum BO, Hodges LF, Ready D, Graap K, Alarcon RD. Virtual reality exposure therapy for Vietnam veterans with posttraumatic stress disorder. J Clin Psychiatry. 2001 Aug;62(8):617-22. doi: 10.4088/jcp.v62n0808. PMID 11561934
- [Background] Difede J, Cukor J, Jayasinghe N, Patt I, Jedel S, Spielman L, Giosan C, Hoffman HG. Virtual reality exposure therapy for the treatment of posttraumatic stress disorder following September 11, 2001. J Clin Psychiatry. 2007 Nov;68(11):1639-47. PMID 18052556
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Koenen KC, Stellman JM, Stellman SD, Sommer JF Jr. Risk factors for course of posttraumatic stress disorder among Vietnam veterans: a 14-year follow-up of American Legionnaires. J Consult Clin Psychol. 2003 Dec;71(6):980-6. doi: 10.1037/0022-006X.71.6.980. PMID 14622073
- [Background] Simms LJ, Watson D, Doebbeling BN. Confirmatory factor analyses of posttraumatic stress symptoms in deployed and nondeployed veterans of the Gulf War. J Abnorm Psychol. 2002 Nov;111(4):637-47. doi: 10.1037//0021-843x.111.4.637. PMID 12428777
- [Background] Hoge CW, Auchterlonie JL, Milliken CS. Mental health problems, use of mental health services, and attrition from military service after returning from deployment to Iraq or Afghanistan. JAMA. 2006 Mar 1;295(9):1023-32. doi: 10.1001/jama.295.9.1023. PMID 16507803
- [Background] Seal KH, Bertenthal D, Miner CR, Sen S, Marmar C. Bringing the war back home: mental health disorders among 103,788 US veterans returning from Iraq and Afghanistan seen at Department of Veterans Affairs facilities. Arch Intern Med. 2007 Mar 12;167(5):476-82. doi: 10.1001/archinte.167.5.476. PMID 17353495
- [Background] Bryant RA. Cognitive behavior therapy of violence-related posttraumatic stress disorder. Aggression and Violent Behavior. 2000;5:79-97.
- [Background] Bryant RA, Moulds ML, Guthrie RM, Dang ST, Nixon RD. Imaginal exposure alone and imaginal exposure with cognitive restructuring in treatment of posttraumatic stress disorder. J Consult Clin Psychol. 2003 Aug;71(4):706-12. doi: 10.1037/0022-006x.71.4.706. PMID 12924676
- [Background] Foa EB. Psychosocial treatment of posttraumatic stress disorder. J Clin Psychiatry. 2000;61 Suppl 5:43-8; discussion 49-51. PMID 10761678
- [Background] Foa EB, Rothbaum BO. Treating the Trauma of Rape: Cognitive-behavioral Therapy for PTSD. New York: Guilford Press; 1998.
- [Background] Foa EB, Meadows EA. Psychosocial treatments for posttraumatic stress disorder: a critical review. Annu Rev Psychol. 1997;48:449-80. doi: 10.1146/annurev.psych.48.1.449. PMID 9046566
- [Background] Carlson JG, Chemtob CM, Rusnak K, Hedlund NL, Muraoka MY. Eye movement desensitization and reprocessing (EDMR) treatment for combat-related posttraumatic stress disorder. J Trauma Stress. 1998 Jan;11(1):3-24. doi: 10.1023/A:1024448814268. PMID 9479673
- [Background] Sherman JJ. Effects of psychotherapeutic treatments for PTSD: a meta-analysis of controlled clinical trials. J Trauma Stress. 1998 Jul;11(3):413-35. doi: 10.1023/A:1024444410595. PMID 9690185
- [Background] Van Etten ML, Taylor S. Comparative efficacy of treatments for Post-traumatic Stress Disorder: A meta-analysis. Clinical Psychology and Psychotherapy. 1998;5:126-144.
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003388. doi: 10.1002/14651858.CD003388.pub2. PMID 15846661
- [Background] Resick PA, Nishith P, Weaver TL, Astin MC, Feuer CA. A comparison of cognitive-processing therapy with prolonged exposure and a waiting condition for the treatment of chronic posttraumatic stress disorder in female rape victims. J Consult Clin Psychol. 2002 Aug;70(4):867-79. doi: 10.1037//0022-006x.70.4.867. PMID 12182270
- [Background] Rothbaum BO, Meadows EA, Resick P, Foy D. Cognitive-behavioral therapy. In: Foa EB, Keane TM, Friedman MJ, eds. Effective Treatments for PTSD: Practice Guidelines from the International Society for Traumatic Stress Studies. New York: Guilford Press; 2000:320-325.
- [Background] Foa EB, Kozak MJ. Emotional processing of fear: exposure to corrective information. Psychol Bull. 1986 Jan;99(1):20-35. No abstract available. PMID 2871574
- [Background] Foa EB, Steketee GS, Rothbaum BO. Behavioral/cognitive conceptualizations of post-traumatic stress disorder. Behavior Therapy. 1989;20:155-176.
- [Background] Foa EB, Hearst-Ikeda D. Emotional Dissociation in Response to Trauma: An Information-Processing Approach. In: Michelson LK, Ray WJ, eds. Handbook of Dissociation: Theoretical and Clinical Perspectives. New York: Plenum Press; 1996:207-222.
- [Background] Delahanty DL, Raimonde AJ, Spoonster E. Initial posttraumatic urinary cortisol levels predict subsequent PTSD symptoms in motor vehicle accident victims. Biol Psychiatry. 2000 Nov 1;48(9):940-7. doi: 10.1016/s0006-3223(00)00896-9. PMID 11074232
- [Background] Shalev AY, Sahar T, Freedman S, Peri T, Glick N, Brandes D, Orr SP, Pitman RK. A prospective study of heart rate response following trauma and the subsequent development of posttraumatic stress disorder. Arch Gen Psychiatry. 1998 Jun;55(6):553-9. doi: 10.1001/archpsyc.55.6.553. PMID 9633675
- [Background] Mason J, Southwick S, Yehuda R, Wang S, Riney S, Bremner D, Johnson D, Lubin H, Blake D, Zhou G, et al. Elevation of serum free triiodothyronine, total triiodothyronine, thyroxine-binding globulin, and total thyroxine levels in combat-related posttraumatic stress disorder. Arch Gen Psychiatry. 1994 Aug;51(8):629-41. doi: 10.1001/archpsyc.1994.03950080041006. PMID 8042912
- [Background] Yehuda R. Post-traumatic stress disorder. N Engl J Med. 2002 Jan 10;346(2):108-14. doi: 10.1056/NEJMra012941. No abstract available. PMID 11784878
- [Background] Yehuda R, Siever LJ, Teicher MH, Levengood RA, Gerber DK, Schmeidler J, Yang RK. Plasma norepinephrine and 3-methoxy-4-hydroxyphenylglycol concentrations and severity of depression in combat posttraumatic stress disorder and major depressive disorder. Biol Psychiatry. 1998 Jul 1;44(1):56-63. doi: 10.1016/s0006-3223(98)80007-3. PMID 9646884
- [Background] Morgan CA 3rd, Grillon C, Southwick SM, Davis M, Charney DS. Exaggerated acoustic startle reflex in Gulf War veterans with posttraumatic stress disorder. Am J Psychiatry. 1996 Jan;153(1):64-8. doi: 10.1176/ajp.153.1.64. PMID 8540594
- [Background] Shalev AY, Peri T, Orr SP, Bonne O, Pitman RK. Auditory startle responses in help-seeking trauma survivors. Psychiatry Res. 1997 Mar 3;69(1):1-7. doi: 10.1016/s0165-1781(96)03001-6. PMID 9080539
- [Background] Lating JM, Everly GS, Jr. Psychophysiological assessment of PTSD. In: Everly, GS, Jr., Lating LM, eds. Psychotraumatology: Key papers and core concepts in post-traumatic stress. New York: Plenum Press; 1995:129-145.
- [Background] Malloy PF, Fairbank JA, Keane TM. Validation of a multimethod assessment of posttraumatic stress disorders in Vietnam veterans. J Consult Clin Psychol. 1983 Aug;51(4):488-94. doi: 10.1037//0022-006x.51.4.488. No abstract available. PMID 6619355
- [Background] Orr SP, Lasko NB, Shalev AY, Pitman RK. Physiologic responses to loud tones in Vietnam veterans with posttraumatic stress disorder. J Abnorm Psychol. 1995 Feb;104(1):75-82. doi: 10.1037//0021-843x.104.1.75. PMID 7897056
- [Background] Pitman RK, Orr SP, Altman B, Longpre RE, Poire RE, Macklin ML, Michaels MJ, Steketee GS. Emotional processing and outcome of imaginal flooding therapy in Vietnam veterans with chronic posttraumatic stress disorder. Compr Psychiatry. 1996 Nov-Dec;37(6):409-18. doi: 10.1016/s0010-440x(96)90024-3. PMID 8932965
- [Background] Keane TM, Kaloupek DG. Imaginal flooding in the treatment of a posttraumatic stress disorder. J Consult Clin Psychol. 1982 Feb;50(1):138-40. doi: 10.1037//0022-006x.50.1.138. No abstract available. PMID 7056906
- [Background] Boudewyns P, Hyer L. Physiological response to combat memories and preliminary treatment outcome in Vietnam veteran PTSD patients treated with direct therapeutic exposure. Behavior Therapy. 1990;21 (1):63-87.
- [Background] Britt TW. The stigma of psychological problems in a work environment: Evidence from the screening of Service Members returning from Bosnia. J of Applied Psych. 2000;30(8):1599-1618.
- [Background] Cardena E, Spiegel D. Dissociative reactions to the San Francisco Bay Area earthquake of 1989. Am J Psychiatry. 1993 Mar;150(3):474-8. doi: 10.1176/ajp.150.3.474. PMID 8434665
- [Background] Koopman C, Classen C, Spiegel D. Predictors of posttraumatic stress symptoms among survivors of the Oakland/Berkeley, Calif., firestorm. Am J Psychiatry. 1994 Jun;151(6):888-94. doi: 10.1176/ajp.151.6.888. PMID 8184999
- [Background] Foa EB, Riggs DS, Massie ED, Yarczower M. The impact of fear activation and anger on the efficacy of exposure treatment for PTSD. Behavior Therapy. 1995;26:487-499.
- [Background] Reger GM, McGee JS, van der Zaag C, Thiebaux M, Galen Buckwalter JG, Rizzo AA. A 3D virtual environment rod and frame test: the reliability and validity of four traditional scoring methods for older adults. J Clin Exp Neuropsychol. 2003 Dec;25(8):1169-77. doi: 10.1076/jcen.25.8.1169.16733. PMID 14566588
- [Background] Rizzo AA, Buckwalter JG, van der Zaag C. Virtual Environment Applications for Neuropsychological Assessment and Rehabilitation. In: Stanney K, ed. Handbook of Virtual Environments. New York: L.A. Earlbaum; 2002:1027-1064.
- [Background] Rothbaum BO, Hodges L, Watson BA, Kessler CD, Opdyke D. Virtual reality exposure therapy in the treatment of fear of flying: a case report. Behav Res Ther. 1996 May-Jun;34(5-6):477-81. doi: 10.1016/0005-7967(96)00007-1. PMID 8687369
- [Background] Rothbaum BO, Hodges L, Smith S, Lee JH, Price L. A controlled study of virtual reality exposure therapy for the fear of flying. J Consult Clin Psychol. 2000 Dec;68(6):1020-6. doi: 10.1037//0022-006x.68.6.1020. PMID 11142535
- [Background] Rothbaum BO, Hodges L, Anderson PL, Price L, Smith S. Twelve-month follow-up of virtual reality and standard exposure therapies for the fear of flying. J Consult Clin Psychol. 2002 Apr;70(2):428-32. doi: 10.1037//0022-006x.70.2.428. PMID 11952201
- [Background] Smith SG, Rothbaum BO, Hodges L. Treatment of fear of flying using virtual reality exposure therapy: A single case study. The Behavior Therapist. 1999;22(8):154-158,160.
- [Background] Rothbaum BO, Hodges LF, Kooper R, Opdyke D, Williford JS, North M. Effectiveness of computer-generated (virtual reality) graded exposure in the treatment of acrophobia. Am J Psychiatry. 1995 Apr;152(4):626-8. doi: 10.1176/ajp.152.4.626. PMID 7694917
- [Background] Emmelkamp PM, Krijn M, Hulsbosch AM, de Vries S, Schuemie MJ, van der Mast CA. Virtual reality treatment versus exposure in vivo: a comparative evaluation in acrophobia. Behav Res Ther. 2002 May;40(5):509-16. doi: 10.1016/s0005-7967(01)00023-7. PMID 12038644
- [Background] Anderson P, Rothbaum BO, Hodges LF. Virtual reality exposure in the treatment of social anxiety: Two case reports. Cognitive and Behavioral Practice. 2003;10:240-247.
- [Background] Botella C, Banos RM, Perpina C, Villa H, Alcaniz M, Rey A. Virtual reality treatment of claustrophobia: a case report. Behav Res Ther. 1998 Feb;36(2):239-46. doi: 10.1016/s0005-7967(97)10006-7. PMID 9613029
- [Background] Carlin AS, Hoffman HG, Weghorst S. Virtual reality and tactile augmentation in the treatment of spider phobia: a case report. Behav Res Ther. 1997 Feb;35(2):153-8. doi: 10.1016/s0005-7967(96)00085-x. PMID 9046678
- [Background] Garcia-Palacios A, Hoffman H, Carlin A, Furness TA 3rd, Botella C. Virtual reality in the treatment of spider phobia: a controlled study. Behav Res Ther. 2002 Sep;40(9):983-93. doi: 10.1016/s0005-7967(01)00068-7. PMID 12296495
- [Background] Rothbaum BO, Anderson P, Zimand E, Hodges L, Lang D, Wilson J. Virtual reality exposure therapy and standard (in vivo) exposure therapy in the treatment of fear of flying. Behav Ther. 2006 Mar;37(1):80-90. doi: 10.1016/j.beth.2005.04.004. Epub 2006 Feb 24. PMID 16942963
- [Background] Botella C, Perpina C, Banos RM, Garcia-Palacios A. Virtual reality: a new clinical setting lab. Stud Health Technol Inform. 1998;58:73-81. PMID 10350931
- [Background] Gershon J, Zimand E, Lemos R, Rothbaum BO, Hodges L. Use of virtual reality as a distractor for painful procedures in a patient with pediatric cancer: a case study. Cyberpsychol Behav. 2003 Dec;6(6):657-61. doi: 10.1089/109493103322725450. PMID 14756933
- [Background] Glantz K, Rizzo AA, Graap K. Virtual reality for psychotherapy: Current reality and future possibilities. Psychotherapy: Theory, Research, Practice, Training. 2003;40(1/2):55-67.
- [Background] Rizzo AA, Schultheis MT, Kerns K, Mateer C. Analysis of assets for virtual applications in neuropsychology. Neuropsychological Rehabilitation. 2004;14(1/2):207-239.
- [Background] Rizzo AA, Kim G. A SWOT analysis of the field of virtual reality and therapy. Presence: Teleoperators and Virtual Environments. 2005;14(2):1-28.
- [Background] Rizzo AA, Rothbaum BO, Graap K. Virtual Reality Applications for Combat-Related Posttraumatic Stress Disorder. In: Figley CR, Nash WP, eds. For Those Who Bore the Battle: Combat Stress Injury Theory, Research, and Management. New York: Taylor and Francis Books; 2006.
- [Background] Rothbaum BO, Hodges L, Alarcon R, Ready D, Shahar F, Graap K, Pair J, Hebert P, Gotz D, Wills B, Baltzell D. Virtual reality exposure therapy for PTSD Vietnam Veterans: a case study. J Trauma Stress. 1999 Apr;12(2):263-71. doi: 10.1023/A:1024772308758. PMID 10378165
- [Background] Rothbaum BO, Ruef AM, Litz BT, Han H, Hodges L. Virtual reality exposure therapy of combat-related PTSD: A case study using psychophysiological indicators of outcome. Journal of Cognitive Psychotherapy. 2003;17(2):163-177.
- [Background] Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. Am J Psychiatry. 2005 Feb;162(2):214-27. doi: 10.1176/appi.ajp.162.2.214. PMID 15677582
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences. Hillsdale: Lawrence Earlbaum Associates; 1988.
- [Background] Cohen J, Cohen P. Applied Multiple Regression/Correlation Analysis for the Behavioral Sciences. Hillsdale: Lawrence Earlbaum; 1983.
- [Background] Foa EB, Hembree E, Rothbaum BO. Prolonged Exposure Therapy for PTSD: Emotional Processing of Traumatic Experiences. New York: Oxford University Press; 2007.
- [Background] Nishith P, Resick PA. Adherence and competence rating scales for prolonged exposure treatment: Unpublished Rating Scale, University of Missouri-St. Louis; 1994.
- [Background] Blake DD, Weathers FW, Nagy LM, Kaloupek DG, Gusman FD, Charney DS, Keane TM. The development of a Clinician-Administered PTSD Scale. J Trauma Stress. 1995 Jan;8(1):75-90. doi: 10.1007/BF02105408. PMID 7712061
- [Background] Schnurr PP, Friedman MJ, Foy DW, Shea MT, Hsieh FY, Lavori PW, Glynn SM, Wattenberg M, Bernardy NC. Randomized trial of trauma-focused group therapy for posttraumatic stress disorder: results from a department of veterans affairs cooperative study. Arch Gen Psychiatry. 2003 May;60(5):481-9. doi: 10.1001/archpsyc.60.5.481. PMID 12742869
- [Background] Aziz MA, Kenford S. Comparability of telephone and face-to-face interviews in assessing patients with posttraumatic stress disorder. J Psychiatr Pract. 2004 Sep;10(5):307-13. doi: 10.1097/00131746-200409000-00004. PMID 15361745
- [Background] Blanchard EB, Jones-Alexander J, Buckley TC, Forneris CA. Psychometric properties of the PTSD Checklist (PCL). Behav Res Ther. 1996 Aug;34(8):669-73. doi: 10.1016/0005-7967(96)00033-2. PMID 8870294
- [Background] Bolton EE, Gray MJ, Litz BT. A cross-lagged analysis of the relationship between symptoms of PTSD and retrospective reports of exposure. J Anxiety Disord. 2006;20(7):877-95. doi: 10.1016/j.janxdis.2006.01.009. Epub 2006 Mar 10. PMID 16530379
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Mackenzie CS, Knox VJ, Gekoski WL, Macaulay HL. An adaptation and extension of the Attitudes Toward Seeking Professional Psychological Help scale. J of Applied Psych. 2004;34(11):2410-2435.
- [Background] Mackenzie CS, Gekoski WL, Knox VJ. Age, gender, and the underutilization of mental health services: the influence of help-seeking attitudes. Aging Ment Health. 2006 Nov;10(6):574-82. doi: 10.1080/13607860600641200. PMID 17050086
- [Background] Ajzen I. From intentions to actions: A theory of planned behavior. In: Kuhl J, Beckman, J, eds. Action-Control: From Cognition to Behavior. Heidelberg: Springer; 1985:11-39.
- [Background] Komiya N, Good GE, Sherrod NB. Emotional openness as a predictor of college students' attitudes toward seeking psychological help. J Counsel Psychol. 2000;47(1):138-143.
- [Background] Pyne JM, Kuc EJ, Schroeder PJ, Fortney JC, Edlund M, Sullivan G. Relationship between perceived stigma and depression severity. J Nerv Ment Dis. 2004 Apr;192(4):278-83. doi: 10.1097/01.nmd.0000120886.39886.a3. PMID 15060401
- [Background] Kennedy RS, Lane NE, Berbaum KS, Lilienthal MG. Simulator Sickness Questionnaire: An enhanced method for quantifying simulator sickness. International Journal of Aviation Psychology. 1993;3(3):203-220.
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Derived] Bourassa KJ, Stevens ES, Katz AC, Rothbaum BO, Reger GM, Norr AM. The Impact of Exposure Therapy on Resting Heart Rate and Heart Rate Reactivity Among Active-Duty Soldiers With Posttraumatic Stress Disorder. Psychosom Med. 2020 Jan;82(1):108-114. doi: 10.1097/PSY.0000000000000758. PMID 31880749